CLINICAL TRIAL: NCT00845000
Title: Acute Effects of SCH 420814 on Dyskinesia and Parkinsonism in Levodopa Treated Patients
Brief Title: Acute Effects of Preladenant (SCH 420814) on Dyskinesia and Parkinsonism in Levodopa Treated Participants (P05550)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P05550; MK-3814-023 (Other: Merck Study Number)
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Results first posted 2016-07-21 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — 2-(2-furanyl)-7-(2-(4-(4-(2-methoxyethoxy)phenyl)-1-piperazinyl)ethyl)-7H-pyrazolo(4,3-e)(1,2,4)triazolo(1,5-c)pyrimidine-5-amine; Levodopa; Carbidopa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- SCH 420814 10 mg→SCH 420814 100 mg→Placebo (Experimental): Participants were to receive their assigned experimental treatment based on randomly assigned treatment sequence at Hour 0 following an overnight withdrawal of their antiparkinsonian medications of each treatment period. The levodopa infusion was to be started at Hour 1 and was to run for 2 hours. The participants were to also receive 25 mg of carbidopa at the following times: Hours 0, 2, and 4. Treatment periods were to be separated by at least 7 days but not more than 28 days washout between each dose.
  Interventions: Drug: SCH 420814 10 mg; Drug: SCH 420814 100 mg; Drug: Placebo; Drug: Levodopa; Drug: Carbidopa
- SCH 420814 100 mg→Placebo→ SCH 420814 10 mg (Experimental): Participants were to receive their assigned experimental treatment based on randomly assigned treatment sequence at Hour 0 following an overnight withdrawal of their antiparkinsonian medications of each treatment period. The levodopa infusion was to be started at Hour 1 and was to run for 2 hours. The participants were to also receive 25 mg of carbidopa at the following times: Hours 0, 2, and 4. Treatment periods were to be separated by at least 7 days but not more than 28 days washout between each dose.
  Interventions: Drug: SCH 420814 10 mg; Drug: SCH 420814 100 mg; Drug: Placebo; Drug: Levodopa; Drug: Carbidopa
- Placebo→SCH 420814 10 mg→SCH 420814 100 mg (Experimental): Participants were to receive their assigned experimental treatment based on randomly assigned treatment sequence at Hour 0 following an overnight withdrawal of their antiparkinsonian medications of each treatment period. The levodopa infusion was to be started at Hour 1 and was to run for 2 hours. The participants were to also receive 25 mg of carbidopa at the following times: Hours 0, 2, and 4. Treatment periods were to be separated by at least 7 days but not more than 28 days washout between each dose.
  Interventions: Drug: SCH 420814 10 mg; Drug: SCH 420814 100 mg; Drug: Placebo; Drug: Levodopa; Drug: Carbidopa
- SCH 420814 10 mg→ Placebo→ SCH 420814 100 mg (Experimental): Participants were to receive their assigned experimental treatment based on randomly assigned treatment sequence at Hour 0 following an overnight withdrawal of their antiparkinsonian medications of each treatment period. The levodopa infusion was to be started at Hour 1 and was to run for 2 hours. The participants were to also receive 25 mg of carbidopa at the following times: Hours 0, 2, and 4. Treatment periods were to be separated by at least 7 days but not more than 28 days washout between each dose.
  Interventions: Drug: SCH 420814 10 mg; Drug: SCH 420814 100 mg; Drug: Placebo; Drug: Levodopa; Drug: Carbidopa
- SCH 420814 100 mg→ SCH 420814 10 mg→Placebo (Experimental): Participants were to receive their assigned experimental treatment based on randomly assigned treatment sequence at Hour 0 following an overnight withdrawal of their antiparkinsonian medications of each treatment period. The levodopa infusion was to be started at Hour 1 and was to run for 2 hours. The participants were to also receive 25 mg of carbidopa at the following times: Hours 0, 2, and 4. Treatment periods were to be separated by at least 7 days but not more than 28 days washout between each dose.
  Interventions: Drug: SCH 420814 10 mg; Drug: SCH 420814 100 mg; Drug: Placebo; Drug: Levodopa; Drug: Carbidopa
- Placebo→ SCH 420814 100 mg→SCH 420814 10 mg (Experimental): Participants were to receive their assigned experimental treatment based on randomly assigned treatment sequence at Hour 0 following an overnight withdrawal of their antiparkinsonian medications of each treatment period. The levodopa infusion was to be started at Hour 1 and was to run for 2 hours. The participants were to also receive 25 mg of carbidopa at the following times: Hours 0, 2, and 4. Treatment periods were to be separated by at least 7 days but not more than 28 days washout between each dose.
  Interventions: Drug: SCH 420814 10 mg; Drug: SCH 420814 100 mg; Drug: Placebo; Drug: Levodopa; Drug: Carbidopa

INTERVENTIONS:
Drug: SCH 420814 10 mg — one 10-mg capsule, orally, at hour 0 of treatment period
Drug: SCH 420814 100 mg — single oral dose of four SCH 420814 25-mg capsules at hour 0 of treatment period
Drug: Placebo — Placebo capsule, oral, at hour 0 of treatment period
Drug: Levodopa — levodopa intravenous (IV) infusion (1 mg/kg body weight) was beginning 1 hour after study drug administration and continued for 2 hours
Drug: Carbidopa — one 25-mg table, orally, at hours 0, 2 and 4 of each treatment period

SUMMARY:
This is a randomized, placebo-controlled, 3-period crossover, balanced, single-site, third party-blind study of preladenant (SCH 420814) in participants with Parkinson disease (PD) to be conducted in conformance with Good Clinical Practices. This trial will investigate the effects of single doses of preladenant and placebo on the dyskinesia and antiparkinsonian actions of a levodopa infusion. The study will examine 10 mg ("low dose") or 100 mg ("high dose") study drug, given as single, oral administrations in conjunction with intravenous (IV) levodopa infusion and oral carbidopa.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have a diagnosis of idiopathic PD based on history, exam and any relevant laboratory tests
* Participants must have been treated with levodopa for one or more years
* Participants must have motor fluctuations that can be measured as a 10% change in tapping speed between "on" and "off" and concurrent motor Unified PD Rating Scale (UPDRS) must also show a 20% improvement when "on"
* Participants must have dyskinesia when "on" measured as at least 2 in one or more body parts on scale using 0 (absent) to 4 (severe) for four limbs, trunk, neck and face (total 7 body parts and 28 points)
* Participant must be free of any clinically significant disease that would interfere with the study evaluations
* Female participants must be postmenopausal and/or surgically sterilized and have a negative serum pregnancy test at the screening visit and a negative urine or serum pregnancy test upon each admission to the study center
* Premenopausal, unsterilized female participants have to agree to use a medically accepted method of contraception
* Male participants must agree to use a medically accepted method of contraception as or abstain from sexual intercourse during the trial and for 2 months after stopping the medication.

Exclusion Criteria:

* Female participants who are pregnant, intend to become pregnant (within 3 months of ending the study), or are lactating
* Participants with dementia (mini-mental state examination [MMSE] <23), hallucinations, confusion, major psychiatric disorders, and unstable medical conditions
* Participants with any stable surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of any drug
* Participants with a positive screen for drugs of abuse
* Participants who are positive for hepatitis B surface antigen, hepatitis C antibodies or human immunodeficiency virus (HIV)
* Participants who are currently participating in another medical interventional clinical study or have participated in a medical interventional clinical study within 30 days and who have previously received this compound.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-04-21 (Actual); Primary Completion 2010-04-30 (Actual); Study Completion 2010-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Period: Period 1
Arm/Group | SCH 420814 10 mg→SCH 420814 100 mg→Placebo | SCH 420814 100 mg→Placebo→ SCH 420814 10 mg | Placebo→SCH 420814 10 mg→SCH 420814 100 mg | SCH 420814 10 mg→ Placebo→ SCH 420814 100 mg | SCH 420814 100 mg→ SCH 420814 10 mg→Placebo | Placebo→ SCH 420814 100 mg→SCH 420814 10 mg
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | SCH 420814 10 mg→SCH 420814 100 mg→Placebo | SCH 420814 100 mg→Placebo→ SCH 420814 10 mg | Placebo→SCH 420814 10 mg→SCH 420814 100 mg | SCH 420814 10 mg→ Placebo→ SCH 420814 100 mg | SCH 420814 100 mg→ SCH 420814 10 mg→Placebo | Placebo→ SCH 420814 100 mg→SCH 420814 10 mg
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | SCH 420814 10 mg→SCH 420814 100 mg→Placebo | SCH 420814 100 mg→Placebo→ SCH 420814 10 mg | Placebo→SCH 420814 10 mg→SCH 420814 100 mg | SCH 420814 10 mg→ Placebo→ SCH 420814 100 mg | SCH 420814 100 mg→ SCH 420814 10 mg→Placebo | Placebo→ SCH 420814 100 mg→SCH 420814 10 mg
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SCH 420814 10 mg→SCH 420814 100 mg→Placebo | SCH 420814 100 mg→Placebo→ SCH 420814 10 mg | Placebo→SCH 420814 10 mg→SCH 420814 100 mg | SCH 420814 10 mg→ Placebo→ SCH 420814 100 mg | SCH 420814 100 mg→ SCH 420814 10 mg→Placebo | Placebo→ SCH 420814 100 mg→SCH 420814 10 mg | Total
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.5 (4.9) | 59.5 (3.5) | 65.0 (4.2) | 63.5 (6.4) | 68.5 (13.4) | 57.5 (3.5) | 61.9 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 2 | 2 | 1 | 6
  Male | 2 | 2 | 1 | 0 | 0 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Mean Peak Dyskinesia Score
Description: Dyskinesia was scored on a scale of 0 (absent), 1 (mild) , 2 (moderate), 3 (severe) and 4 (incapacitating) for seven body parts (face, neck, trunk, each arm and each leg) based on the worse dyskinesia noted during the entire measurement time. Scores were assessed at Hours 0, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 7.0 and 8.0. The dyskinesia score was the sum of the scores for the seven body parts. The peak dyskinesia score was recorded for each participant regardless of what timepoint the score was achieved. The total possible score for an individual at each timepoint could range from 0 to 28 with higher scores indicating greater effects of the dyskinesia. The mean peak dyskinesia score was calculated using the individual peak values.
Time Frame: Hours 0, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 7.0 and 8.0 of each treatment period
Population: All participants who received at least 1 dose of study drug and had available data for endpoint. Results pooled by study drug and not by randomly assigned sequence.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- SCH 420814 10 mg: Participants who received single oral dose of SCH 420814 10 mg in either period 1, 2, or 3 regardless of randomly assigned treatment sequence
- SCH 420814 100 mg: Participants who received single oral dose of SCH 420814 100 mg (four 25 mg capsules) in either period 1, 2, or 3 regardless of randomly assigned treatment
- Placebo: Participants who received placebo in either period 1, 2, or 3 regardless of randomly assigned treatment
Arm/Group | SCH 420814 10 mg | SCH 420814 100 mg | Placebo
Number analyzed (Participants) | 12 | 12 | 12
Score on a scale | 11.00 (5.15) | 11.42 (5.81) | 8.50 (3.92)

2. Secondary Outcome: Mean Peak Finger Tapping Score
Description: Tapping was measured with two manual counters with keys that were depressed to register a count. The participant alternately tapped each counter using the index finger of the more affected hand for 60 seconds and was not allowed to use more than one finger to tap. The participant was instructed to tap as rapidly as possible while being timed for 60 seconds. The counts were recorded for the two counters at Hours 0, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 7.0 and 8.0. The peak tapping score was recorded for each participant regardless of what timepoint the score was achieved. The mean peak finger tapping score was calculated using the individual peak values.
Time Frame: Hours 0, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 7.0 and 8.0 of each treatment period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: taps per 60 seconds
Arm/Group | SCH 420814 10 mg | SCH 420814 100 mg | Placebo
Number analyzed (Participants) | 12 | 12 | 12
taps per 60 seconds | 44.33 (27.76) | 41.58 (22.31) | 45.75 (28.26)

3. Secondary Outcome: Mean Peak Tremor Score
Description: Tremor was scored on a scale of 0 (absent), 1 (mild, 2 (moderate), 3 (severe) and 4 (incapacitating) for seven body parts (face, neck, trunk, each arm and each leg) based on the worse tremor observed during the time spent with participant while taking other study measurements(vital signs, drawing samples, performing the tapping and walking tasks). Scores were assessed at Hours 0, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 7.0 and 8.0. The tremor score was the sum of scores for seven body parts. The peak tremor score was recorded for each participant regardless of what timepoint the score was achieved. The total possible score for an individual at each timepoint could range from 0 to 28 with higher scores indicating more effects of the tremors. The mean peak tremor score was calculated using the individual peak values.
Time Frame: Hours 0, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 7.0 and 8.0 of each treatment period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | SCH 420814 10 mg | SCH 420814 100 mg | Placebo
Number analyzed (Participants) | 12 | 12 | 12
Score on a scale | 3.5 (4.76) | 3.33 (4.66) | 4.42 (5.30)

4. Secondary Outcome: Mean Peak Walking Speed
Description: Walking speed assessment began with the participant being seated in an armless chair. Then while being timed, the participant stood up with their arms crossed on their chest and walked 6 meters, turned around, returned to the chair and sat. Timing was stopped when the participant's buttocks hit the chair and the total time was recorded. If the participant could not arise in 60 seconds, 60 seconds was entered in this line of the report form and the participant was tested again but allowed to push off to get out of the chair. Sixty seconds was the maximum time allowed to complete the walking assessment, thus 60 seconds was recorded as the time if they could not complete the task within this time limit. Walking speed was assessed at Hours 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 7.0 and 8. The peak walking speed was recorded for each participant regardless of what timepoint the score was achieved. The mean peak walking speed was calculated using the individual peak values.
Time Frame: Hours 0, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 7.0 and 8.0 of each treatment period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | SCH 420814 10 mg | SCH 420814 100 mg | Placebo
Number analyzed (Participants) | 12 | 12 | 12
Seconds | 16.64 (18.98) | 14.45 (15.73) | 20.00 (20.64)

ADVERSE EVENTS:
Time Frame: up to 70 days (up to 14 days after last dose of study drug)
Description: Safety population included all participants who received at least 1 dose of study drug. Adverse events are reported by study drug administered at time of the event and not by randomly assigned sequence.
Groups:
- Placebo: Participants who received single oral dose of placebo in either period 1, 2, or 3 regardless of randomly assigned treatment
Arm/Group | SCH 420814 10 mg | SCH 420814 100 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 5/12 | 4/12 | 4/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCH 420814 10 mg (N=12) | SCH 420814 100 mg (N=12) | Placebo (N=12)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
INFUSION SITE EXTRAVASATION (General disorders) | 0 (0) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
THERMAL BURN (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
ATAXIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
DYSKINESIA (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
DYSTONIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 4 (6) | 2 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish or publicly present any interim results of the trial without the prior written consent of the sponsor. The investigator further agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the trial.